CLINICAL TRIAL: NCT06505720
Title: Arthroscopic Versus Open Management of Acute Pediatric Septic Hip Infection: A Randomized Controlled Trial
Brief Title: Use of Arthroscopy in Treatment of Acute Pediatric Septic Hip Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hesham Mohamed Elbaseet (Other)
Responsible Party: Sponsor-Investigator, Hesham Mohamed Elbaseet, MD, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ٍSeptic Hip in childern
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acute Pediatric Septic Hip Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The child in this group will be treated for his\ her acute septic hip infection using open surgery ( The Standard Method)
  Interventions: Procedure: Open debridement of acute pediatric septic hip
- Intervention Group (Other): The child in this group will be treated for his\ her acute septic hip infection arthroscopically
  Interventions: Procedure: Arthroscopic management of acute pediatric septic hip infecion

INTERVENTIONS:
Procedure: Arthroscopic management of acute pediatric septic hip infecion — Three-portals tractionless hip arthroscopy will be used to treat acute pediatric septic hip infection
  Arms: Intervention Group
Procedure: Open debridement of acute pediatric septic hip — surgical drainage and debridement of acute septic hip in children via classic lateral approach
  Arms: Control Group

SUMMARY:
Acute septic hip infection in pediatric population is a true orthopedic surgical emergency that require early diagnosis and prompt management. Open surgical debridement and drainage of the hip through lateral approach is the gold standard method of treatment. Usage of hip arthroscopy in the treatment of such condition has been in clinical practice for more than 30 years. However, literature is still lacking in actual prospective comparison about the outcome of both methods.

DETAILED DESCRIPTION:
The study will divide the children presented with acute septic hip infection into two groups; the control group in which the child will undergo traditional open surgical debridement and drainage of the hip via lateral approach, and the intervention group in which arthroscopic drainage and debridement of the hip will be done. The outcomes of both methods will be recorded and compared. The research hypothesis is that arthroscopic management of acute pediatric septic hip infection is as effective as open surgery; with fewer complications and faster recovery.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 months - 14 years _unilateral or bilateral acute septic hip arthritis

Exclusion Criteria:

* Children with pre-existing other pathology of the affected hip, whether he / she has surgery for management of this pathology or not.

  * Patients whose parents refuse to participate in the study

Ages: 10 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2024-08-13 (Estimated); Primary Completion 2026-02-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Modified Mckay's criteria | One Year Follow-up
  Excellent: painless, stable hip; no limp; more than 15 degrees of internal rotation.
  Good: painless, stable hip; slight limb or decreased motion , negative Trendelenburg sign Fair: minimum pain; moderate stiffness, positive Trendelenburg sign Poor: significant pain.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fabry G, Meire E. Septic arthritis of the hip in children: poor results after late and inadequate treatment. J Pediatr Orthop. 1983 Sep;3(4):461-6. doi: 10.1097/01241398-198309000-00008. PMID 6630490
- [Background] Sucato DJ, Schwend RM, Gillespie R. Septic Arthritis of the Hip in Children. J Am Acad Orthop Surg. 1997 Oct;5(5):249-260. doi: 10.5435/00124635-199709000-00003. PMID 10795061
- [Background] Kocher MS, Mandiga R, Zurakowski D, Barnewolt C, Kasser JR. Validation of a clinical prediction rule for the differentiation between septic arthritis and transient synovitis of the hip in children. J Bone Joint Surg Am. 2004 Aug;86(8):1629-35. doi: 10.2106/00004623-200408000-00005. PMID 15292409
- [Background] Shaw BA, Kasser JR. Acute septic arthritis in infancy and childhood. Clin Orthop Relat Res. 1990 Aug;(257):212-25. PMID 2199119
- [Background] DeAngelis NA, Busconi BD. Hip arthroscopy in the pediatric population. Clin Orthop Relat Res. 2003 Jan;(406):60-3. doi: 10.1097/01.blo.0000043044.84315.90. PMID 12579000
- [Background] Ellis HB, Copley L, Pennock A, Nepple JJ, Willimon C, Mayer SW, Yen YM. Tractionless Hip Arthroscopy for Septic Arthritis in Children. Arthrosc Tech. 2021 Feb 19;10(3):e659-e667. doi: 10.1016/j.eats.2020.10.079. eCollection 2021 Mar. PMID 33738199
- [Background] El-Sayed AM. Treatment of early septic arthritis of the hip in children: comparison of results of open arthrotomy versus arthroscopic drainage. J Child Orthop. 2008 Jun;2(3):229-37. doi: 10.1007/s11832-008-0094-0. Epub 2008 Mar 6. PMID 19308583
- [Background] Bennett OM, Namnyak SS. Acute septic arthritis of the hip joint in infancy and childhood. Clin Orthop Relat Res. 1992 Aug;(281):123-32. PMID 1499198
- [Background] Donders CM, Spaans AJ, Bessems JHJM, van Bergen CJA. A systematic review of the optimal drainage technique for septic hip arthritis in children. Hip Int. 2022 Sep;32(5):685-693. doi: 10.1177/1120700021989666. Epub 2021 Feb 10. PMID 33566696
- [Background] McKay DW. A comparison of the innominate and the pericapsular osteotomy in the treatment of congenital dislocation of the hip. Clin Orthop Relat Res. 1974 Jan-Feb;(98):124-32. doi: 10.1097/00003086-197401000-00013. No abstract available. PMID 4817221